CLINICAL TRIAL: NCT00076791
Title: A Phase I Study of the Safety, Tolerance, and Pharmacokinetics of Tenofovir Disoproxil Fumarate (TDF) and the Combination of TDF Plus Emtricitabine in HIV-1 Infected Pregnant Women and Their Infants
Brief Title: Safety of Tenofovir Disoproxil Fumarate (TDF) and Emtricitabine/TDF in HIV Infected Pregnant Women and Their Infants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); International Maternal Pediatric Adolescent AIDS Clinical Trials Group (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P394; 10034 (Registry Identifier: DAIDS ES); PACTG 394; IMPAACT 394
Record Dates: First submitted 2004-02-03; First posted 2004-02-06 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: HIV Seronegativity
MeSH Terms: conditions — HIV Infections | interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Tenofovir

ARMS (2):
- 1 (Active Comparator): Each participant in Cohort 1 received a single 600 mg oral dose of TDF at the start of active labor or 4 hours prior to C-section, with concurrent administration of standard intravenous zidovudine (ZDV) prophylaxis and/or other antiretrovirals prescribed by her physician. The infants from Cohort 1 received only the standard 6 weeks of oral ZDV prophylaxis postpartum.
  Interventions: Drug: Emtricitabine/Tenofovir disoproxil fumarate; Drug: Tenofovir disoproxil fumarate
- 2 (Active Comparator): Mothers in Cohort 2 will receive a single dose of 900 mg of TDF combined with 600 mg emtricitabine, along with standard ZDV prophylaxis and/or other antiretrovirals prescribed by her physician. Infants will receive a single dose of TDF at 4 mg/kg combined with 3 mg/kg emtricitabine as soon as possible after delivery and within 6 hours of age as well as the standard 6 weeks of oral ZDV prophylaxis after birth.
  Interventions: Drug: Emtricitabine/Tenofovir disoproxil fumarate; Drug: Tenofovir disoproxil fumarate

INTERVENTIONS:
Drug: Emtricitabine/Tenofovir disoproxil fumarate — 900 mg of TDF combined with 600 mg emtricitabine
Drug: Tenofovir disoproxil fumarate — 600 mg oral dose of TDF

SUMMARY:
Most infants infected with HIV through mother-to-child transmission (MTCT, or perinatal transmission) become infected during labor and delivery. The purpose of this study is to test the safety and tolerability of a single dose of tenofovir disoproxil fumarate (TDF) or emtricitabine/TDF (FTC/TDF) given at the time of labor to HIV infected pregnant women and to their newborn infants.

DETAILED DESCRIPTION:
The majority of perinatally infected infants are infected during the labor and delivery process, but recent studies suggest that additional factors, such as postexposure prophylaxis, are likely to be involved in the prevention of MTCT of HIV. It is possible that antiretroviral dosing only during labor and short-term dosing to newly born infants would be sufficiently effective to prevent MTCT of HIV. TDF is a nucleoside reverse transcriptase inhibitor that has demonstrated significant effectiveness in preventing MTCT of simian immunodeficiency virus (SIV) in a primate model of HIV. FTC/TDF is a combination of two NRTIs being studied because this combination has the potential to prevent MTCT, while protecting the mother from developing resistance that may develop with single drug therapy. This study will evaluate the safety, tolerance, and pharmacokinetics (PK) of single doses of TDF and FTC/TDF in both HIV infected pregnant women and their newborn infants.

Cohort 1 is now closed. Each participant in Cohort 1 received a single 600 mg oral dose of TDF at the start of active labor or 4 hours prior to C-section, with concurrent administration of standard intravenous zidovudine (ZDV) prophylaxis and/or other antiretrovirals prescribed by her physician. The infants from Cohort 1 received only the standard 6 weeks of oral ZDV prophylaxis postpartum. PK blood samples were taken from mothers at predose and 1, 2, 4, 8, 12, and 24 hours postdose and at the time of delivery; PK blood samples were taken from infants at 12, 24, and 36 hours after birth.

Pregnant women with HIV infection entering this study will be assigned to Cohort 2, as all infants in Cohort 1 have completed the 6 to 8 week study visit and all Cohort 1 data have been reviewed. Mothers in Cohort 2 will receive a single dose of 900 mg of TDF combined with 600 mg emtricitabine, along with standard ZDV prophylaxis and/or other antiretrovirals prescribed by her physician. Infants will receive a single dose of TDF at 4 mg/kg combined with 3 mg/kg emtricitabine as soon as possible after delivery and within 6 hours of age as well as the standard 6 weeks of oral ZDV prophylaxis after birth. Blood samples from mothers and infants will be taken as for Cohort 1.

Mothers will be followed for 12 weeks postpartum or for 2 years after giving birth if viral resistance to TDF or FTC/TDF is demonstrated at Weeks 1, 6, or 12. In addition to the PK studies, blood collection will occur around the time of delivery, at screening, study entry, at delivery, and after delivery at various times up to Week 12. Physical exams will be done at screening, study entry, at delivery, and after delivery at various times up to Week 8. Infants will be followed until age 2. Blood will be collected and physical exams will be done at birth and at various times up to Week 96. Mothers are encouraged to coenroll in PACTG P1025, Pharmacokinetic Study of Anti-HIV Drugs During Pregnancy.

ELIGIBILITY:
Inclusion Criteria for Mothers:

* HIV infected
* 34 weeks or more (third trimester) into pregnancy at study screening
* Have access to a participating AIDS clinical trial unit (ACTU) and are willing to be followed at location for the duration of the study

Exclusion Criteria for Mothers:

* Prior treatment with TDF, including coformulated drugs that contain TDF, during current pregnancy
* Active opportunistic infection and/or serious bacterial infection at time of study entry
* Certain abnormal laboratory values at study screening
* Chronic malabsorption or chronic diarrhea
* Certain medical or obstetrical complications during the current pregnancy
* Fetal abnormalities as measured by ultrasound screening performed at 18 weeks into pregnancy or later
* Intend to breastfeed
* Current alcohol abuse or use of illicit substances
* Participation in any other therapeutic or vaccine perinatal treatment trial during the current pregnancy, unless given permission by the protocol chairs
* Require certain medications

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2004-03; Primary Completion 2010-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Adverse experiences with a severity of Grade 3 or 4 and adverse pregnancy outcomes that cannot be directly attributed to a cause besides study treatment | Throughout study

SECONDARY OUTCOMES:
Maternal viral load | during active labor and 24 to 48 hours, 7 days, 6 to 8 weeks, and 12 weeks postpartum
viral resistance to emtricitabine/tenofovir disoproxil fumarate using bulk sequencing | at Weeks 1, 6, and 12 postpartum
infant HIV DNA PCR | at 24 to 48 hours, 6 to 8 weeks, 4 months, and 6 months of life

CONTACTS AND LOCATIONS:
Overall Officials: Patricia M. Flynn, MD, Study Chair — Department of Infectious Disease, St. Jude's Children's Research Hospital; Arlene D. Bardeguez, MD, MPH, FACOG, Study Chair — Obstetrics, Gynecology, and Women's Health, University of Medicine and Dentistry of New Jersey
Locations (12):
- United States (11):
  - Children's National Med. Ctr. Washington DC NICHD CRS, Washington D.C., District of Columbia
  - Washington Hosp. Ctr. NICHD CRS, Washington D.C., District of Columbia
  - Univ. of Miami Ped. Perinatal HIV/AIDS CRS, Miami, Florida
  - Mt. Sinai Hosp. Med. Ctr. - Chicago, Womens & Childrens HIV Program, Chicago, Illinois
  - Children's Hospital of Michigan NICHD CRS, Detroit, Michigan
  - NJ Med. School CRS, Newark, New Jersey
  - Nyu Ny Nichd Crs, New York, New York
  - Bronx-Lebanon Hosp. IMPAACT CRS, The Bronx, New York
  - Hahnemann Univ. Hosp., Philadelphia, Pennsylvania
  - Regional Med. Ctr. at Memphis, Memphis, Tennessee
  - St. Jude/UTHSC CRS, Memphis, Tennessee
- San Juan City Hosp. PR NICHD CRS, San Juan, Puerto Rico

REFERENCES:
- [Background] Antoniou T, Park-Wyllie LY, Tseng AL. Tenofovir: a nucleotide analog for the management of human immunodeficiency virus infection. Pharmacotherapy. 2003 Jan;23(1):29-43. doi: 10.1592/phco.23.1.29.31915. PMID 12523458
- [Background] Kourtis AP, Duerr A. Prevention of perinatal HIV transmission: a review of novel strategies. Expert Opin Investig Drugs. 2003 Sep;12(9):1535-44. doi: 10.1517/13543784.12.9.1535. PMID 12943497
- [Background] Moodley J, Moodley D. Management of human immunodeficiency virus infection in pregnancy. Best Pract Res Clin Obstet Gynaecol. 2005 Apr;19(2):169-83. doi: 10.1016/j.bpobgyn.2004.10.007. Epub 2004 Dec 15. PMID 15778108
- [Background] Abrams EJ. Prevention of mother-to-child transmission of HIV--successes, controversies and critical questions. AIDS Rev. 2004 Jul-Sep;6(3):131-43. PMID 15595430
- [Background] Thorne C, Newell ML. The safety of antiretroviral drugs in pregnancy. Expert Opin Drug Saf. 2005 Mar;4(2):323-35. doi: 10.1517/14740338.4.2.323. PMID 15794723